CLINICAL TRIAL: NCT03755440
Title: Phase II Study of PD-1 Antibody SHR-1210 in EBV Positive Metastatic Gastric Cancer Patients.
Brief Title: PD-1 Antibody in EBV Positive Metastatic Gastric Cancer Patients.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Ruihua Xu, Professor, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EBVaGC-SYSUCC
Record Dates: First submitted 2018-11-22; First posted 2018-11-28 (Actual); Last update posted 2022-09-21 (Actual); Status verified 2022-09

CONDITIONS: Gastric Cancer Stage IV; EBV
Keywords: EBV; Gatric cancer; Check point inhibitor
MeSH Terms: conditions — Stomach Neoplasms | interventions — camrelizumab

STUDY DESIGN:
Intervention Model Description: PD-1 antibody, SHR-1210
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PD-1 antibody (Experimental): SHR-1210, 200mg, ivdrip, d1, every two weeks.
  Interventions: Drug: PD-1 antibody (SHR-1210)

INTERVENTIONS:
Drug: PD-1 antibody (SHR-1210) — PD-1 antibody (SHR-1210), 200mg, ivdrip, every 2 weeks.

SUMMARY:
EBV positive tumor accounts for 8-9% of all gastric cancer (GC) patients. PD-1 antibody has been proved as third line therapy for PD-L1 positive gastric cancer. Previous studies showed that EBV(+) tumors exhibit high response to PD-1 antibody. In this phase II study, we will investigate the efficacy and safety of PD-1 antibody in EBV positive metastatic GC patients.

DETAILED DESCRIPTION:
EBV positive metastatic GC patients who failed to standard chemotherapy will receive therapy of single agent, PD-1 antibody, SHR-1210, 200mg, every 2 weeks. The primary endpoint is response rate. Secondary endpoint is progress free survival, overall survival, safety and quality of life. Using the Simon two-stage sample size calculation, the sample size is 19. We will collect tissue and blood sample for exploratory analysis, including PD-L1 stuatus, tumor mutation burden, et al.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed Recurrent/Metastatic gastric adenocarcinoma;
2. EBER positive;
3. Failed from first-line platinum and fluorouracil based chemotherapy and second-line chemotherapy; or could not tolerate systematic chemotherapy
4. ECOG performance status of 0 or 1;
5. Life expectancy ≥ 12 weeks;
6. Subjects must have measurable disease by CT or MRI per RECIST 1.1 criteria;
7. Can provide either a newly obtained or archival tumor tissue sample;
8. Adequate laboratory parameters during the screening period as evidenced by the following:

   Absolute neutrophil count ≥ 1.5 × 10^9/L ; Platelets ≥ 90 × 10^9/L; Hemoglobin ≥ 9.0 g/dL; Serum albumin ≥ 2.8g/dL; Total bilirubin (TBIL) ≤ 1.5 × upper limit of normal (ULN), ALT and AST ≤ 1.5×ULN Creatinine clearance≥50 mL/min;
9. Female of child bearing potential, a negative urine or serum pregnancy test result within 72 h before study treatment. Participants of reproductive potential must be willing to use adequate contraception for the course of the study through 60 days after the last dose of SHR-1210. Male subjects must be willing to use adequate contraception for the course of the study through 120 days after the last dose of SHR-1210;
10. Subjects must be willing to participate in the research and sign an informed consent form (ICF);

Exclusion Criteria:

1. Subjects with any active autoimmune disease or history of autoimmune disease;
2. Subjects having clinical symptoms of metastases to central nervous system (such as cerebral edema, requiring steroids intervention, or brain metastasis progression);
3. Has a known additional malignancy within the last 5 years before study treatment with the exception of curatively treated basal cell and squamous cell carcinoma of the skin and/or curatively resected in-situ cervical cancers;
4. Uncontrolled clinically significant heart disease, including but not limited to the following: (1) > NYHA II congestive heart failure; (2) unstable angina, (3) myocardial infarction within the past 1 year; (4) clinically significant supraventricular arrhythmia or ventricular arrhythmia requirement for treatment or intervention;
5. Concurrent medical condition requiring the use of cortisol (>10mg/day Prednisone or equivalent dose) or other systematic immunosuppressive medications within 14 days before the study treatment. Except: inhalation or topical corticosteroids. Doses > 10 mg/day prednisone or equivalent for replacement therapy;
6. Has received prior anti-cancer monoclonal antibody (mAb), chemotherapy, targeted small molecule therapy within 4 weeks prior to first dosing or not recovered to ≤CTCAE 1 from adverse events (except for hair loss or neurotoxic sequelae from prior platinum therapy) due to a previously administered agent. 7. Palliative irradiation finished within 2 weeks;

8. Active infection or an unexplained fever > 38.5°C before two weeks of first dosing (subjects with tumor fever may be enrolled at the discretion of the investigator); 9. Known Human Immunodeficiency Virus (HIV) infection、active Hepatitis B or Hepatitis C; 10. Currently participating or has participated in a study within 4 weeks of the first dose of study medication; 11. Pregnancy or breast feeding; 12. Prior therapy with a PD-1, anti-PD-Ligand 1 (PD-L1) or CTLA-4 agent; 13. Subjects are known to have a history of psychiatric substance abuse, alcoholism, or drug addiction; 14. According to the investigator, other conditions that may lead to stop the research.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2018-12-01 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Response rate | From first patient first visit to 6 month after last patient first visit ] Based on Response Evaluation Criteria in Solid Tumors 1.1 (RECIST 1.1)
  The percentage of patients whose cancer shrinks or disappears after treatment

SECONDARY OUTCOMES:
Progression-Free Survival (PFS) | up to approximately 1 year
  PFS as measured in accordance with the Response Evaluation Criteria In Solid Tumours (RECIST) version 1.1
Overall Survival (OS) | up to approximately 2 year
  The time from registration to death due to any cause, or censored at date last known alive.
Disease Control Rate (DCR) | From first patient first visit to 6 month after last patient first visit
  Based on Response Evaluation Criteria in Solid Tumors 1.1 (RECIST 1.1)

CONTACTS AND LOCATIONS:
Overall Officials: Rui-Hua Xu, MD, PhD, Principal Investigator — Sun Yat-sen University
Locations (1):
- Cancer center of Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Sun YT, Guan WL, Zhao Q, Wang DS, Lu SX, He CY, Chen SZ, Wang FH, Li YH, Zhou ZW, Xu RH, Qiu MZ. PD-1 antibody camrelizumab for Epstein-Barr virus-positive metastatic gastric cancer: a single-arm, open-label, phase 2 trial. Am J Cancer Res. 2021 Oct 15;11(10):5006-5015. eCollection 2021. PMID 34765307